CLINICAL TRIAL: NCT06643741
Title: Collection of Pregnancy Outcome Data and Whole Blood Samples From Women Undergoing Non-Invasive Screening for Early, Preterm, and Term Preeclampsia
Brief Title: Non-Invasive Preeclampsia Screening and Biobank
Status: Recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Rutgers Robert Wood Johnson Medical School (Other); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-PRE-401
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia (PE)
Keywords: preeclampsia; pregnant
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Whole blood processed to plasma and serum will be obtained from all subjects. A subset of subjects will be asked to provide remnant placental tissue following delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant subjects between 11 and 14 weeks gestation.: This is an observational study and no study-specific intervention is defined. PE screen test results will not be reported back to the physician or subject but will be compared to birth outcome data.

SUMMARY:
Women pregnant between 11-14 weeks gestation will be enrolled with blood samples collected to evaluate for preeclampsia.

DETAILED DESCRIPTION:
To collect relevant pregnancy outcome data, medical history, and blood samples from pregnant women carrying a singleton fetus undergoing non-invasive screening for early, preterm and term pre-eclampsia (PE) starting at 11 weeks 0 days to 14 weeks 0 days (≥11 - ≤14) gestation in support of validating the Labcorp Preeclampsia ScreenTM assay. Data will be used to examine assay performance and develop new testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female and 18 years of age and older;
* Subject provides a signed and dated informed consent;
* Subject is pregnant with a singleton pregnancy at ≥11.0 - ≤14.0 weeks' gestation;
* Subject agrees to provide the Sponsor access to any prenatal and postnatal screening or diagnostic test results and supporting data;
* Subject agrees to have UtAPI calculated during their SOC first trimester ultrasound and MAP collected at the first trimester SOC visit;
* Subject agrees to provide up to 25mL of whole blood at each trimester visit;
* Subject agrees to provide relevant medical and pregnancy/postnatal information including outcome.

Exclusion Criteria:

* Subject is unlikely to return for second and third trimester testing;
* Subject is unlikely to have pregnancy outcome data available;
* Previous sample donation under this protocol with the same pregnancy;
* Subject is participating in a blinded aspirin study or taking unknown doses of aspirin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject is pregnant with a singleton pregnancy at ≥11.0 - ≤14.0 weeks' gestation
Sampling Method: Non-Probability Sample
Enrollment: 6550 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Baseline serum samples will be used to evaluate the performance of the Labcorp Preeclampsia Screen assay | From enrollment at 10-14 weeks gestation until pregnancy outcome is available, up to 36 weeks
  The results of the Preeclampsia Screen assay will be compared to pregnancy outcome data to evaluate how well the assay predicted early onset PE (<34 weeks gestational age) and preterm PE (<37 weeks gestational age).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosenfeld, DO, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (21):
- United States (21):
  - Valley Perinatal, Glendale, Arizona
  - Delaware Center for Maternal and Fetal Medicine, Newark, Delaware
  - D&H National Research Centers, Miami, Florida
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cooper University Health Care, Camden, New Jersey
  - New Jersey Perinatal Associates, Livingston, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Capital Health, Pennington, New Jersey
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - St. David's Women's Center of Texas, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UT Health, Houston, Texas
  - HCA Healthcare, Texas Maternal Fetal Medicine, Houston, Texas
  - Macon & Joan Brock Virginia Health Sciences at Old Dominion University, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No